CLINICAL TRIAL: NCT05244083
Title: Effectiveness of the Mirror Therapy for Improving Bimanual Performance, Somatosensory Function of the Impaired Upper Limb and Quality of Life in Children With Unilateral Spastic Cerebral Palsy: A Randomised Clinical Trial
Brief Title: Effectiveness of the Mirror Therapy for Improving Bimanual Performance, Somatosensory Function of the Impaired Upper Limb and Quality of Life in Children With Unilateral Spastic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Anna Ortega I Martínez, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIS-2021-07
Record Dates: First submitted 2022-01-07; First posted 2022-02-17 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Hemiplegic Cerebral Palsy; Mirror Movement Therapy
Keywords: unilateral spastic cerebral palsy; mirror therapy; bimanual performance; somatosensory function; quality of life
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will perform a 5-week motor program consisting of 4 bimanual exercises with mirror therapy, to be done at home 30 minutes a day, 5 days a week.
  Interventions: Other: Mirror Therapy
- Control Group (Active Comparator): The control group will perform a 5-week motor program consisting of 4 bimanual exercises without mirror therapy, to be done at home 30 minutes a day, 5 days a week.
  Interventions: Other: Program without Mirror Therapy

INTERVENTIONS:
Other: Mirror Therapy — Therapy consisting of perfoming bimanual activities with a mirror placed on the patient's sagital plane, so it creates the brain illusion that the impaired limb moves the same way and quality that the unimpaired does.
  Arms: Experimental Group
Other: Program without Mirror Therapy — Bimanual exercises performed with both upper limbs.
  Arms: Control Group

SUMMARY:
* Background: Unilateral Spastic Cerebral Palsy (USPC) is caused by an injury in one brain hemisphere in the immature brain, and affects the contralateral side of the body, especially on the upper limb. It induces motor and somatosensory damages, that are closely related to the hand function. Evidence posits mirror therapy to be a therapy with potential effects on bimanual performance and somatosensory function, that may influence on quality of life. The aim of this study is to demonstrate the effectiveness of a motor program with mirror therapy in children with USCP in the improvement of the bimanual performance, the somatosensory function and quality of life compared with the same program without mirror.
* Methods: This study is a Randomised Clinical Trial. The participants are children with USCP aged between 8 and 12 years old classified in levels I and II in Manual Ability Classification System, recruited from Fundació Aspace Catalunya. The eligibility criteria are a) to not have had surgical interventions, botulinum toxin or shock waves 3 months before the study; b) to not be receiving intensive therapies on the upper limb; c) to not have attentional or behavioural difficulties; d) to not have moderate to high intellectual disability; e) to not have non-treated epilepsy; and f) to not have non-corrected visual problems. A total of 22 participants will be recruited for this study, and will be randomised in two groups: control and experimental, through the opaque envelope technique. The experimental group will perform a 5-week motor program consisting of 4 bimanual exercises with mirror therapy, to be done at home 30 minutes a day, 5 days a week, while the control group will perform the same program without the mirror. The assessments will be done by a blinded evaluator and will include bimanual performance (Children's Hand-use Experience Questionnaire), somatosensory function and quality of life (PedsQL™), and will be performed at the beginning, at the end of the intervention and 1-month follow-up.
* Discussion: Favourably results in this study may imply the implementation of a low-cost therapy, suitable to be done at home, and with no contraindications for children with USCP. Moreover, the suitability to be adapted and performed at home could increase the family implication and empowerment, increasing its confidence in the disability process.

ELIGIBILITY:
Inclusion Criteria:

* To have been diagnosed with Unilateral Spastic Cerebral Palsy.
* To be capable of following and understanding rules.

Exclusion Criteria:

* To have had surgical interventions, botulinum toxin or shock waves 3 months before the study;
* To be receiving intensive therapies on the upper limb;
* To have attentional or behavioural difficulties;
* To have moderate to high intellectual disability;
* To have non-treated epilepsy;
* To have non-corrected visual problems

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Bimanual Performance | Baseline, at 5 weeks and at 9 weeks
  How Bimanual Performance, assessed with Children's Hand-use Experience Questionnaire, changes by doing the intervention

SECONDARY OUTCOMES:
Change in Tactile Registration of the impaired hand. | Baseline, at 5 weeks and at 9 weeks
  An evaluation to determine whether the impaired hand is capable of identifying a somatosensory stimuli. The index pad is stimulated with the Semmes Weinstein Monofilament, starting with the largest monofilament considered as "normal sensation. 3 correct identifications are considered as a correct answer, with the smallest monofilament possible.
Change in static two-point discrimination of the impaired hand. | Baseline, at 5 weeks and at 9 weeks
  An evaluation to determine the shortest distance that the impaired hand is capable of identifying to simultaneous stimuli.The index pad is stimulated with the Disk-Criminator, that applies two simultaneous stimuly. The shortest distance at which the patient is capable of idenitfying both stimuli 7/10 times is considered as a correct answer.
Change in moving two-point discrimination of the impaired hand. | Baseline, at 5 weeks and at 9 weeks
  An evaluation to determine the shortest distance that the impaired hand is capable of identifying to moving simultaneous stimuli.The index pad is stimulated with the Disk-Criminator, that applies two simultaneous stimuly, with small circular movement. The shortest distance at which the patient is capable of idenitfying both stimuli 7/10 times is considered as a correct answer.
Change in single point localisation of the impaired hand. | Baseline, at 5 weeks and at 9 weeks
  An evaluation to determine both the capacity of the patient to identify a threshold stimuly applied to thumb, index, 4th and 5th finger of the impaired hand, and the position where stimuli is applied (front, back or side). 12 different stimulations are applied, and the correct answers are the final punctuation.
Change in double simultaneous of the impaired hand. | Baseline, at 5 weeks and at 9 weeks
  An evaluation to determine the capacity of the patient to identify a threshold stimuly applied to thumb, index, 4th and 5th finger of the impaired hand, and on the same fingers of the other hand, single and combined. 24 different stimulations are applied, and the correct answers are the final punctuation.
Change in sterognosis of the impaired hand. | Baseline, at 5 weeks and at 9 weeks
  An evaluation to determine the capacity of the patient to identify 9 different objects (pen, pencil, button, coin, safety pin, paper clip, key, peg and spoon) placed on the impaired hand, without visual feedback. The final punctuation is for the correct identifications.
Self-reported Quality of Life | Baseline, at 5 weeks and at 9 weeks
  How the self-perceived quality of life, assessed with Pediatric Quality of Life Inventory (PEDSQL - CP Module), changes by performing the intervention. The evaluation consists of gradinf (from 0 - never; to 4 - always), how have different situations caused trouble or impairment to children. The presented situations are related to daily activities, movement, pain, school activities, comunication, feeding and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA CARITAT BAGUR CALAFAT, PHD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Fundació Aspace Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes